## Assessing the Clinical Performance of Two Frequent Replacement Silicone Hydrogel Multifocal Contact Lenses

STUDY ID

CLN705-M102

**PROTOCOL** 

NCT05702541



# Feasibility Clinical Protocol for CLN705-M102 Title: Assessing the Clinical Performance of Two Frequent Replacement Silicone Hydrogel Multifocal Contact Lenses

| Protocol Number and Version: | CLN705-M102, Version 4.0 |
|---|---|
| Sponsor Name and | Alcon Research, LLC and its affiliates ("Alcon") |
| Address: | 6201 South Freeway Fort Worth, Texas 76134-2099 |
| Test Product(s): | LID223194 MF SiHy Contact lenses |

#### **Sponsor Contact Details**



Property of Alcon
Confidential
May not be used, divulged, published, or otherwise disclosed without the consent of
Alcon

Document ID: V-CLN-0035558

Status: Approved, Version: 4.0  Approved Date: 11 Jan 2023

Investigator Agreement:

- I have read the Feasibility Clinical Protocol described herein and the Feasibility Clinical Master Protocol governing it, recognize its confidentiality, and agree to conduct the described trial in compliance with Good Clinical Practice (GCP), the ethical principles contained within the Declaration of Helsinki, this protocol, all applicable regulatory authority regulations, and conditions of approval imposed by the reviewing IRB or regulatory authority.
- I will supervise all testing of the device involving human subjects and ensure that the requirements relating to obtaining informed consent and IRB review and approval are met in accordance with applicable local and governmental regulations.
- I have read and understand the appropriate use of the investigational product(s) as described in the protocol, current Investigator's Brochure, product information, or other sources provided by the sponsor.
- I understand the potential risks and side effects of the investigational product(s).
- I agree to maintain adequate and accurate records in accordance with government regulations and to make those records available for inspection.
- I agree to comply with all other requirements regarding the obligations of clinical investigators and all other pertinent requirements of the sponsor and government agencies.
- I agree to ensure that all associates, colleagues, and employees assisting in the conduct of the study are informed of their obligations in meeting the above commitments.

| | Have you ever been disqualified as an investigator by any Regulatory Authoric □ No □Yes | ty? |
|---|---|---|
| | Have you ever been involved in a study or other research that was terminated? □ No □ Yes | |
| | If yes, please explain here: | |
| Pr | cipal investigator | |
| | Signature Date 1 | te |
| | ne and professional ition: | |
| Αc | lress: | |

## **Table of Contents**

| Feasibility ( | Clinical Protocol for CLN705-M102 | 1 |
|---------------|----------------------------------------------|------------|
| Table of Co | ontents | 3 |
| List of Tabl | les | 3 |
| Abbreviatio | ons and Acronyms | 4 |
| | BILITY CLINICAL PROTOCOL | |
| 1.2 | Study Overview | |
| 1.3 | Study Product and Associated Materials | 13 |
| 1.4 | Study-Specific Lens Returns | 19 |
| | 1.4.1 Worn IP | 19 |
| | 1.4.2 Lens Return (ADE/Device Deficiency) | 19 |
| | List of Tables | |
| Table 1-1 | Schedule of Study Procedures and Assessments | 1 <i>6</i> |

## **Abbreviations and Acronyms**

| Abbreviation | Definition |
|--------------|----------------------------------------------|
| ADE | Adverse device effect |
| AE | Adverse event |
| BCVA | Best corrected visual acuity |
| °C | Degrees Celsius |
| CDMA | Clinical Development & Medical Affairs |
| CSS | Clinical Site Specialist |
| CT&OL | Clinical Trial & Operations Lead |
| D | Diopter(s) |
| eCRF | Electronic case report form |
| GA | Georgia |
| GCP | Good Clinical Practice |
| ICF | Informed consent form |
| ID | Identification |
| IP | Investigational product |
| IRB | Institutional review board |
| JCR | Johns Creek Research |
| LID | Lens identification number |
| logMAR | Logarithm of the minimum angle of resolution |
| MR | Manifest refraction |
| OD | Right eye |
| OS | Left eye |
| OU | Both eyes |
| PI | Principal investigator |
| R&D | Research & Development |
| SADE | Serious adverse device effect |
| SiHy | Silicone hydrogel |
| US or USA | United States |

| Abbreviation | Definition |
|--------------|---------------|
| VA | Visual acuity |

## 1 FEASIBILITY CLINICAL PROTOCOL



## 1.2 Study Overview

| Protocol Study Details | |
|---|---|
| Study Rationale and Objective | In this clinical trial, clinical performance of LID#223194 Multifocal contact lens and a commercially available Air Optix plus HydraGlyde Multifocal contact lens will be assessed. |
| Investigator(s) Site | Johns Creek Research Clinic<br>11460 Johns Creek Parkway |
| Site | Johns Creek, GA, 30097 USA |
| External Organizations | Not Applicable |
| Planned Duration of Exposure | ~ 4 days total (test and comparator) Test Product (LID223194): 2 days (+ 3 days) Comparator Product (AirOptix HydraGlyde MF [AOHG MF]): 2 days (+3 days) Exposure of study lenses in 2 different periods over 3 visits |
| <b>Number of Subjects</b> | |
| Study Population | <ul> <li>Habitual soft Multifocal contact lens wearers aged ≥ 40 years with normal eyes (not needing ocular medication, other than correction for refractive error). Subjects should have at least 3 months wearing experience, wear these lenses at least 5 days per week and at least 8 hours per day.</li> <li>To qualify, subjects must require cylindrical correction ≤ 0.75D, be able wear study contact lens with sphere power ranging between +3.00D and -7.00D and requiring a near ADD of LO, MED or HI</li> </ul> |
| Lens Assignment | Subjects will be randomized in a 1:1 manner to receive one of 2 lens sequences: |
| | Sequence 1: LID223194/AOHG MF |
| | • Sequence 2: AOHG MF/LID223194 |

| <b>Protocol Study</b> | tudy Details | |
|---|---|---|
| Study Design | □ Prospective | Single-masked (trial subject) |
| | Randomized | Open-label |
| | Single group | Contralateral |
| | Parallel group | |
| | Crossover | Monocular lens wear |
| | Other | |
| | Visit Schedule: | |
| | 1. Visit 1 - Screening/Baseli | - |
| | | Visit 1) Follow-up (to occur at least ion) Lens Pair 1/Dispense Lens 2 |
| | | Visit 2) Follow-up (to occur at least |
| _ | 4-6 hours after lens insert | |
| <b>Decision Criteria</b> | Not applicable | |
| Assessments | 1. VA with study lenses (logMAR; OU) @ 4m | |
| Safety Assessments | 1. AEs | |
| | <ul><li>2. Biomicroscopy</li><li>3. Device deficiencies</li></ul> | |
| | 3. Device deficiencies | |

#### **Protocol Study Details**

#### **Inclusion Criteria**

- 1. Subject must be at least 40 years of age.
- 2. Subject must be able to understand and must sign an informed consent form (ICF) that has been approved by an Institutional Review Board (IRB).
- 3. Subject must be willing to stop wearing their habitual contact lenses for the duration of study participation.
- 4. Currently wears multifocal soft contact lenses in both eyes for a minimum of 5 days per week and 8 hours per day during the past 3 months.
- 5. Manifest cylinder  $\leq 0.75$  D in each eye.
- 6. BCVA 0.1 logMAR or better in each eye.
- 7. Able to fit with available contact lenses: within a range of powers from +3.00D to -7.00 and requiring a near ADD of LO, MED or HI
- 8. Subject must possess spectacles that provide a corrected visual acuity of 20/40 or better OU

#### **Exclusion Criteria**

- 1. Any anterior segment infection, inflammation, or abnormality or disease (including systemic) that contraindicates contact lens wear, as determined by the investigator.
- 2. Any use of systemic or ocular medications for which contact lens wear could be contraindicated, as determined by the investigator.
- 3. History of refractive surgery or plan to have refractive surgery during the study or irregular cornea in either eye.
- 4. Ocular or intraocular surgery (excluding placement of punctal plugs) within the previous 12 months or planned during the study.
- 5. Biomicroscopy findings at screening that are moderate (Grade 3) or higher and/or corneal vascularization that is mild (Grade 2) or higher, and/or any infiltrate.
- 6. Current or history of pathologically dry eye in either eye that, in the opinion of the investigator, would preclude contact lens wear.
- 7. Current or history of herpetic keratitis in either eye.
- 8. Eye injury in either eye within 12 weeks immediately prior to enrollment for this trial.
- 9. Current or history of intolerance, hypersensitivity, or allergy to any component of the study products.
- 10. The investigator, his/her staff, family members of the investigator, family members of the investigator's staff, or individuals living in the households of the aforementioned persons in the study.

| <b>Protocol Study</b> | Protocol Study Details |
|---|---|
| | <ul><li>11. Participation of the subject in a clinical trial within the previous</li><li>3 days or currently enrolled in any clinical trial.</li><li>12. Monovision contact lens wearer</li></ul> |
| Enrollment<br>Stopping Criteria | Enrollment stopping criteria will not be defined for this study. |

| | Analysis Plan |
|---|---|
| Statistical Analysis | The following product or lens naming conventions will be used: • LID223194 • AOHG MF |
| Subject Characteristics and Study Conduct Summaries | The following will be presented: • Demographics Characteristics (listing) |
| Assessment<br>Analysis Strategy | Results from selected assessment will be summarized using descriptive statistics according to its measurement scale. Listings will be provided as necessary. The Safety Analysis Set will serve as the analysis data set for all effectiveness analyses. |





## 1.3 Study Product and Associated Materials

| | Test Product LID223194 | Comparator Product AIR OPTIX plus HydraGlyde Multifocal |
|---|---|---|
| Primary<br>component/<br>material | Lehfilcon A | Lotrafilcon B |
| Manufactu<br>rer | Alcon Laboratories, Inc. | Alcon Laboratories, Inc. |
| Power<br>Range | <ul> <li>LO Add with +1.00 to -5.00D (in 0.25D steps) spherical power as available</li> <li>MED Add with +3.00D to -7.00D (in 0.25D steps) spherical power as available</li> <li>HI Add with +3.00D to -7.00D (in 0.25D steps) spherical power as available</li> </ul> | <ul> <li>LO Add with +1.00 to -5.00D (in 0.25D steps) spherical power as available</li> <li>MED Add with +3.00D to -7.00D (in 0.25D steps) spherical power as available</li> <li>HI Add with +3.00D to -7.00D (in 0.25D steps) spherical power as available</li> </ul> |
| Supply | The sponsor will provide this test product. | The site will procure this comparator product |

| | Test Product | Comparator Product |
|---|---|---|
| | LID223194 | AIR OPTIX plus HydraGlyde Multifocal |
| Packaging and | Primary label on blister foil pack includes, at a minimum: | Commercial primary label on blister foil pack |
| Labeling | material name or identifier | |
| | base curve | |
| | diameter | |
| | <ul> <li>packing solution</li> </ul> | |
| | • power | |
| | • lot number | |
| | expiration date | |
| | • content statement | |
| | <ul> <li>investigational device statement</li> </ul> | |
| | <ul> <li>sponsor information</li> </ul> | |
| | country of origin | |
| | Secondary color-coded label on packages includes: | |
| | <ul> <li>clinical protocol number</li> </ul> | |
| | <ul> <li>material name or identifier</li> </ul> | |
| | • power | |
| | <ul> <li>an investigational use only statement</li> </ul> | |
| | <ul> <li>tracking or handling unit number</li> </ul> | |
| Storage | Lenses should be stored at room temperature. | Refer to manufacturer's instructions |
| Other | Replacement lenses are allowed only if there is a device deficiency (e.g., torn lens) or if the lens falls on the ground and investigator wants to insert a new lens. | Replacement lenses are allowed only if there is a device deficiency (e.g., torn lens) or if the lens falls on the ground and investigator wants to insert a new lens. |


| | Test Product LID223194 | Comparator Product AIR OPTIX plus HydraGlyde Multifocal |
|---|---|---|
| Associated Materials | <ul> <li>CLEAR CARE Cleaning and Disinfecting Solution will be used with study lenses for the duration of study.</li> <li>LacriPure rinsing/reinsertion PRN will be used as needed with study lenses.</li> <li>Lubrication/re-wetting drops will not be permitted during study lens wear.</li> </ul> | <ul> <li>CLEAR CARE Cleaning and Disinfecting Solution will be used with study lenses for the duration of study.</li> <li>LacriPure rinsing/reinsertion PRN will be used as needed with study lenses.</li> <li>Lubrication/re-wetting drops will not be permitted during study lens wear.</li> </ul> |

 Table 1-1
 Schedule of Study Procedures and Assessments

| | Procedure/ Assessment | Visit 1 | Visit 2 | | Visit 3 | Unscheduled<br>Visit/Early Exit<br>Visit | Source<br>Only* |
|---|---|---|---|---|---|---|---|
| | | Screening/<br>Baseline/<br>Dispense<br>Lens 1 | Follow up Lens 1<br>(2 (+ 3) Days)<br>after Visit 1<br>(minimum 4 -<br>6 hrs after<br>insertion) | Dispense<br>Lens 2 | Follow up Lens 2<br>(2(+3) Days) after<br>Visit 2 (minimum 4-<br>6 hrs after<br>insertion)/Exit | | |
| 1 | Informed Consent | X | | | | | |
| 2 | Demographics | X | | | | | |
| 3 | Medical History | X | X | X | X | X | X |
| 4 | <b>Concomitant Medications</b> | X | X | X | X | X | X |
| 5 | Inclusion/ Exclusion | X | | | | | |
| 6 | Habitual lens<br>(brand, power) | X | | | | | X |
| 7 | VA w/ habitual correction<br>(OD, OS, Snellen distance) | X | (X) | (X) | (X) | (X) | X |
| 8 | Manifest refraction (most plus spherical equivalent) | X | | | | (X) | |
| 9 | BCVA (OD, OS, logMAR; distance and near with manifest refraction) | X | | | | (X) | |
| 10 | Biomicroscopy | X | X | | X | X | |

Document ID: V-CLN-0035558 Status: Approved, Version: 4.0 Approved Date: 11 Jan 2023 

| 13 | Randomize | X | | | | |
|----|------------------------------|---|---|---|---|-----|
| 14 | Dispense study lenses | X | | X | | (X) |
| 18 | VA w/ study lenses, (logMAR) | | | | | |
| | • Distance (4m; OU) | X | X | X | X | (X) |



#### 1.4 Study-Specific Lens Returns

#### 1.4.1 Worn IP

Worn IP will be returned to the sponsor. Use the following instructions for collection, storage, and shipping, unless otherwise instructed by the sponsor.

- Removal from eye: Clean hands
- Storage container: Unused screw-top lens case
- Label information:
  - Protocol number
  - o Site number
  - Subject ID
  - o Eye
  - Lens type/ identification
  - Date collected
- Storage solution: PURILENS Plus Preservative Free Saline (PURILENS Plus Saline)
- Storage temperature: Refrigerated 4-10°C
- Timing of return: Study Completion
- An inventory/list of lenses being returned



Notify via email the CSS and Clinical Trial & Operations Lead when lenses are returned.





